CLINICAL TRIAL: NCT04949269
Title: A Phase 1, Open-label, Crossover Study to Evaluate the Pharmacokinetics of Deucravacitinib (BMS-986165) Administered as Various Solid Tablet Formulations in Healthy Subjects
Brief Title: A Study to Evaluate the Drug Levels of Deucravacitinib From Tablets After Oral Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IM011-120
Record Dates: First submitted 2021-06-30; First posted 2021-07-02 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Deucravacitinib; BMS-986165
MeSH Terms: interventions — deucravacitinib; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental)
  Interventions: Drug: Deucravacitinib
- Part B (Experimental)
  Interventions: Drug: Deucravacitinib
- Part C (Experimental)
  Interventions: Drug: Deucravacitinib; Drug: Famotidine
- Part D (Experimental)
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
Drug: Famotidine — Specified dose on specified days
  Other Names: Pepcid
  Arms: Part C

SUMMARY:
The purpose of this study is to assess the drug levels of deucravacitinib after oral administration in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory determinations.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and total body weight ≥50 kg (110 lb).
* Willing and able to consume 4 units of alcohol (Part C only). Only participants with low to moderate alcohol consumption will be enrolled in Part C of this study (ie, consumption of between 1 and 21 units per week for males and between 1 and 14 units per week in females).

Exclusion Criteria:

* Current or recent (within 3 months or 90 days of study drug administration) clinically significant gastrointestinal disease that, in the opinion of the investigator or medical monitor, could impact upon the absorption of study drug.
* Any medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease.
* Clinically significant history or presence of acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months or 90 days prior to screening.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of deucravacitinib | Up to 7 days
Area Under the Concentration-time Curve from time 0 to 24 hours postdose (AUC(0-24)) of deucravacitinib | Up to 7 days
Concentration at 24 hours of post-morning dose on Day 1 and Day 7 (C24) of deucravacitinib | Up to 7 days

SECONDARY OUTCOMES:
Incidence of non-serious Adverse Events (AEs) | Up to 18 days
Incidence of Serious Adverse Events (SAEs) | Up to 30 days post discontinuation of dosing or participant's participation in the study
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 11 days
Incidence of clinically significant changes in clinical laboratory values: Chemistry tests | Up to 11 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 11 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 11 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 11 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 11 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 11 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 11 days
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in ECG parameters: QRS | Up to 11 days
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in ECG parameters: QT interval | Up to 11 days
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in ECG parameters: QTcF | Up to 11 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Quotient Sciences Miami, Miami, Florida
  - PPD Development, LP, Austin, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html